CLINICAL TRIAL: NCT04021472
Title: Evaluate Health Coaching Support in Technology-based Interventions for Goal Setting (PEC 15-470)
Brief Title: Evaluate Health Coaching Support in Technology-based Interventions for Meeting Health Goals
Acronym: Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PEX 19-002; PEC 15-470 (Other Grant/Funding Number: Office of Connected Care)
Record Dates: First submitted 2019-06-27; First posted 2019-07-16 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Chronic Disease Prevention
Keywords: Disease prevention; Digital health; Text messaging

STUDY DESIGN:
Intervention Model Description: One-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Text message (Experimental): Participants receive text messages about healthy eating or physical activity.
  Interventions: Behavioral: Text message

INTERVENTIONS:
Behavioral: Text message — Two months of daily text messages to support meeting a health goal

SUMMARY:
This was a pilot evaluation conducted to test procedures for a possible future trial and provide preliminary insights regarding whether text messages sent to Veterans could help support nutrition and/or physical activity health goals. For the purposes of the pilot, the goal was to enroll one participant.

DETAILED DESCRIPTION:
The investigators prepared procedures for a one-group pilot intended to evaluate the delivery of automated text messages to Veterans. Completion of this pilot will provide preliminary insights regarding the delivering automated text messages focused on nutrition and/or physical activity health goals, and potential impacts on outcomes like self-efficacy, goal commitment, and health confidence.

ELIGIBILITY:
Inclusion Criteria:

* Patient at designated VA site
* Ownership of a cellular phone
* Over age 18
* Pre-screened by their primary care physician for study inclusion for medical contraindication to physical activity and diet change

Exclusion Criteria:

* Patient outside designated VA site
* Non-ownership of a cellular phone
* Under age 18
* Not pre-screened by their primary care physician for study inclusion for medical contraindication to physical activity and diet change or deemed ineligible to participate by primary care physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Patrick Hogan, PhD MS BS, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Lisa M. Quintiliani, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Text Message
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 81 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Self-efficacy: Healthful Eating Via Revised Eating Self-Efficacy Scale (ESES-R)
Description: Self-reported confidence in performing healthful diet and physical activity behaviors. Self-efficacy - Healthful eating via Revised Eating Self-Efficacy Scale (ESES-R). Range: 1-10; higher values represent a better outcome.
Time Frame: Change from Baseline to 2 months
Measure: Number; unit: score on a scale
Arm/Group | Text Message
Number analyzed (Participants) | 1
score on a scale | 2.3

2. Primary Outcome: Goal Commitment: Healthful Eating Via the Hollenbeck, Williams, and Klein Goal Commitment Scale
Description: Self-reported commitment to healthful diet and physical activity goals. Goal commitment - Healthful eating via the Hollenbeck, Williams, and Klein Goal Commitment Scale. Range: 1-5; higher values represent a better outcome.
Time Frame: Change from Baseline to 2 months
Measure: Number; unit: score on a scale
Arm/Group | Text Message
Number analyzed (Participants) | 1
score on a scale | -0.2

3. Primary Outcome: Self-efficacy: Physical Activity Via the Self-efficacy for Exercise Behaviors Scale
Description: Self-reported confidence in performing healthful diet and physical activity behaviors. Self-efficacy - Physical activity via the Self-efficacy for Exercise Behaviors Scale. Range: 1-5; higher values represent a better outcome.
Time Frame: Change from Baseline to 2 months
Measure: Number; unit: score on a scale
Arm/Group | Text Message
Number analyzed (Participants) | 1
score on a scale | 2.5

4. Primary Outcome: Goal Commitment - Physical Activity Via the Hollenbeck, Williams, and Klein Physical Activity Scale
Description: Self-reported commitment to healthful diet and physical activity goals. The determination to attempt a physical activity-related goal and consistently pursue it over time. Goal commitment - Physical activity via the Hollenbeck, Williams, and Klein Goal Commitment Scale. Range: 1-5; higher values represent a better outcome.
Time Frame: Baseline
Population: This scale was not administered at 2 month follow-up
Measure: Number; unit: score on a scale
Arm/Group | Text Message
Number analyzed (Participants) | 1
score on a scale | 4.2

5. Secondary Outcome: Health Confidence: the Health Confidence Score
Description: Self-reported confidence in patient engagement. Health Confidence. Range: 0-12; higher values represent a better outcome.
Time Frame: Change from Baseline to 2 months
Measure: Number; unit: score on a scale
Arm/Group | Text Message
Number analyzed (Participants) | 1
score on a scale | 0.75

ADVERSE EVENTS:
Time Frame: Data were collected over the course of 3 months.
Arm/Group | Text Message
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04021472/Prot_000.pdf